CLINICAL TRIAL: NCT04296994
Title: A Phase 1, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of QL1706 in Patients With Advanced Malignant Tumor
Brief Title: A Study of QL1706 in Subjects With Advanced Malignant Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-101
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-label Dose Escalation and Expansion Study of QL1706 (Experimental): Part 1 (Dose escalation): QL1706 will be administered in sequential cohorts each receiving 1 of 4 doses of QL1706 on day 1 of every 21-day cycle (3 weeks) via IV infusion. Dose escalation will continue until an MTD is reached.
  Part 2 (Dose Expansion): The PK parameters of QL1706 will be tested at 2-3 doses determined during the dose-escalation phase in subjects with advanced malignant tumor cohorts.
  Interventions: Biological: QL1706

INTERVENTIONS:
Biological: QL1706 — QL1706（PSB205） is a bi-functional product that has been engineered to contain two unique monoclonal antibodies.
  Other Names: PSB205

SUMMARY:
This is an open-label, multicenter, Phase 1, ascending dose escalation study of QL1706 in subjects with advanced malignant tumor. The study will be conducted in 2 parts. Part 1 of the study will be a dose escalation evaluation to determine the maximum tolerated dose (MTD) and to establish a recommended Phase 2 dose (RP2D) of QL1706. This study purpose is to describe the safety and tolerability, to assess Pharmacokinetics (PK) and immunogenicity, and to preliminarily assess the anti-tumor activity of QL1706 in subjects with advanced malignant tumor. Part 2 of the study will further characterize the PK parameters for QL1706 in subjects with advanced malignant tumor.

DETAILED DESCRIPTION:
The study was divided into screening/baseline, treatment and follow-up periods. Safety monitoring will be conducted throughout the study period. DLT will be determined 21 days (1 cycle) after the first administration of QL1706 based on the occurrence of AE during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
3. Life expectancy of ≥3 months.
4. The functional level of important organs must meet the requirements before the first dose of study drug.
5. Male and female patients able to have children must agree to use highly effective method of contraception throughout the study and for at least 180 days after last dose.Female subjects who are not pregnant or breastfeeding.
6. Patients with pathological diagnosis of advanced/metastatic malignant tumor have progressed disease on standard therapy or for which no effective therapy is avalizble.

Exclusion Criteria:

1. Active or prior documented autoimmune disease. Subjects who have stable hypothyroidism with hormone replacement ,childhood atopy or asthma, vitiligo, alopecia, , or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
2. Grade 3 or Grade 4 irAEs related to prior cancer immunotherapy.
3. Known symptomatic brain metastases, leptomeningeal disease or spinal cord compression.
4. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment on decision of investigator. .
5. Any condition requiring systemic treatment with corticosteroids or other immunosuppressive medications within 14 days before first dose of study drug. Corticosteroids for topical use, nasal spray, and inhaled steroids are allowed. Systemic corticosteroids for prophylaxis of contrast allergy are permitted.
6. Systemic anti-cancer treatment. This includes radiotherapy ,small molecule targeted therapy<2 weeks before the first dose of study drug, ≤4 weeks for chemotherapy，monoclonal antibody;≤8 weeks for cell-based therapy or anti-tumor vaccine.
7. Major surgery within 28 days before the first dose of study drug and not recovered fully from any complications from surgery.
8. Systemic infection requiring IV antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
9. Subjects with the history of organ transplant or allogeneic hematopoietic stem cells transpalnt.
10. Positive for Human immunodeficiency virus（HIV）or Hepatitis B ,active Hepatitis C.
11. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 1 Cycles (21 days)
  Safety and tolerability, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Univeisity Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Ma Y, Lin S, Chen Q, Xue J, Yang Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Li W, Li Q, Zhu C, Huang Z, Kang X, Xue S, Li H, Wang C, Luo F, Huang Y, Zhang L, Zhao H. Updated efficacy and predictive biomarkers of QL1706, a bifunctional PD-1/CTLA-4 dual blocker in advanced solid tumors-A phase 1/1b study. Cell Rep Med. 2025 Oct 21;6(10):102396. doi: 10.1016/j.xcrm.2025.102396. Epub 2025 Oct 3. PMID 41045933
- [Derived] Zhao Y, Ma Y, Zang A, Cheng Y, Zhang Y, Wang X, Chen Z, Qu S, He J, Chen C, Jin C, Zhu D, Li Q, Liu X, Su W, Ba Y, Hao Y, Chen J, Zhang G, Qu S, Li Y, Feng W, Yang M, Liu B, Ouyang W, Liang J, Yu Z, Kang X, Xue S, Yang G, Yan W, Yang Y, Liu Z, Peng Y, Fanslow B, Huang X, Zhang L, Zhao H. First-in-human phase I/Ib study of QL1706 (PSB205), a bifunctional PD1/CTLA4 dual blocker, in patients with advanced solid tumors. J Hematol Oncol. 2023 May 8;16(1):50. doi: 10.1186/s13045-023-01445-1. PMID 37158938